CLINICAL TRIAL: NCT03356808
Title: Multicenter Trial of Cancer Antigen-specific T Cells in the Treatment of Lung Cancer
Brief Title: Antigen-specific T Cells Against Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-17023
Record Dates: First submitted 2017-11-24; First posted 2017-11-29 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Lung Cancer
Keywords: Lung cancer; CAR-T; mesothelin; Muc1; GD2; MAGE-A4
MeSH Terms: conditions — Lung Neoplasms; Medullary cystic kidney disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung cancer-specific T cells (Experimental): Peripheral blood mononuclear cells (PBMCs) of patients, who have cancer antigen identified lung cancer, will be obtained through apheresis, and T cells will be activated and ex vivo engineered.
  Interventions: Biological: Lung cancer-specific T cells

INTERVENTIONS:
Biological: Lung cancer-specific T cells — 1 infusion, for 1x10^6~1x10^7 cells/kg via IV

SUMMARY:
The purpose of this clinical trial is to assess the feasibility, safety and efficacy of cancer antigen-specific T cells targeting lung cancer. The cancer targeting antigens are identified through immunostaining of patient's cancer specimens. Another goal of the study is to learn more about the persistence and function of the ex vivo manipulated antigen-specific T cells in the body.

DETAILED DESCRIPTION:
Lung cancer is a malignancy characterized by uncontrolled cell growth in tissues of the lung. There are two main types of lung cancer, small-cell lung carcinoma (SCLC) and non-small-cell lung carcinoma (NSCLC). In 2012, lung cancer occurred in 1.8 million people and resulted in 1.6 million deaths worldwide. Common treatments include surgery, chemotherapy, and radiotherapy, but in relapsed cancer patients, such treatments often have limited successes.

In this study, the participant's peripheral blood mononuclear cells will be collected for antigen-specific T cell preparation, and/or modified using an advanced lentiviral vector system. Then the antigen-specific T cells, called engineered immune effectors (EIEs) or chimeric antigen receptor modified-T cells (CAR T), which can recognize specific molecules that are expressed by the lung cancer cells, are given back to the participant by intravenous infusion.

The purpose of this clinical trial is to assess the feasibility, safety and efficacy of T cell immunotherapy targeting single or multiple cancer antigens. The lung cancer antigens include known tumor antigens such as MAGE-A1, MAGE-A4, MucI, GD2, and mesothelin, as well as novel cancer antigens. Another goal of the study is to learn more about the persistence and function of the specific CAR T cells in the body.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage III, IV or relapsed lung cancer confirmed by histology and biopsy.
2. Age: ≥ 18 years and ≤ 80 years.
3. 4 weeks at least since last chemotherapy or radiotherapy and 2 weeks at least since last systemic steroid hormone and other immunosuppressive therapy.
4. Side Effects of Chemotherapy have subsided.
5. Cancer specific antigens are identified and shown to express at high levels (>2+) in malignant tissues by immuno-histochemical staining or flow cytometry.
6. Karnofsky/Lansky ≥ 50%.
7. Expected survival ≥ 6 weeks.

Initial hematopoietic conditions with

* neutrophils (ANC) ≥ 1×10^6/L;
* platelet (PLT) ≥ 1×10^8/L.

Proper renal and hepatic functions (ULN denotes "upper limit of normal range") with

* serum creatinine ≤ 2×ULN;
* serum bilirubin ≤ 3×ULN;
* AST/ALT ≤ 5×ULN.

  10. Oxygen saturation ≥ 90%. 11. Written, informed consent obtained prior to any study-specific procedures.

Exclusion Criteria:

1. Airway obstruction caused by tumor.
2. History of epilepsy or other central nervous system diseases.
3. Patients who require systemic corticosteroid or other immunosuppressive therapy.
4. History of prolonged or serious heart disease during QT.
5. history of serious cyclophosphamide toxicity.
6. Current or recent treatment (within the 28-day period prior to Day 0) with another investigational drug or previous participation in any immune cell therapy study.

Inadequate liver and renal function with

* serum creatinine > 2.5 mg/dl;
* serum (total) bilirubin > 2.0 mg/dl;
* AST & ALT > 3 x ULN.

  8. Pregnant or lactating females. 9. Serious active infection during screening. 10. Active HIV, Hepatitis B virus (HBV), Hepatitis C virus (HCV) infection or uncontrolled infection.

  11. Patients, in the opinion of investigators, may not be eligible or not able to comply with the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of engineered T cells in patients using CTCAE version 4.0 standard to evaluate the level of adverse events | 3 months
  Physiological parameter (measuring cytokine response)

SECONDARY OUTCOMES:
Persistence and proliferation of engineered antigen-specific T cells in patients | 3 months
  The expansion and functional persistence of ex vivo engineered T cells in the peripheral blood of patients will be examined on Day 7, 14, 21, 28, 60 and 90 after infusion.
Anti-tumor effects | 1 year
  Objective response, such as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) will be assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, PhD, Principal Investigator — Shenzhen Geno-Immune Medical Institute; Qichun Cai, MD, Study Director — Jinshazhou Hospital of Guangzhou University of Chinese Medicine; Xun Lai, MD, Study Director — Yunnan Cancer Hospital & The Third Affiliated Hospital of Kunming Medical University & Yunnan Cancer Center
Locations (3):
- China (3):
  - Jinshazhou Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong
  - Yunnan Cancer Hospital & The Third Affiliated Hospital of Kunming Medical University & Yunnan Cancer Center, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No